CLINICAL TRIAL: NCT04381247
Title: Comprehensive Molecular Diagnosis and Management of Hospital- and Ventilator-associated Pneumonia in Norway
Acronym: HVAPNOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Haukeland University Hospital (Other); University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: VV HVAPNOR
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Pneumonia, Ventilator-Associated; Hospital-acquired Pneumonia; Infectious Disease; Infection, Hospital; Antibiotic Resistant Infection
Keywords: pneumonia; hospital-acquired pneumonia; ventilator-associated pneumonia; molecular diagnostics; biomarker; antibiotic stewardship
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Communicable Diseases; Cross Infection; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Airway sampling, Whole blood, serum, plasma, faecal and urinary samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Molecular diagnostics in HAP and VAP — Airway samples will be analyzed both by standard and molecular based microbiological analysis.

SUMMARY:
HVAPNOR consists of Three work packages:

1. Prospective observational study of Hospital (HAP) - and ventilator-Associated pneumonia (VAP) at 5 hospitals in Norway. Establish optimized routines for microbiological sampling, diagnostics and antibiotic stewardship..
2. Biomarker studies in HAP and VAP.
3. Studies on capacity building in HAP and VAP diagnostics.

DETAILED DESCRIPTION:
Lower respiratory tract infections include hospital-acquired pneumonia (HAP) and ventilator- associated pneumonia (VAP) with a very high mortality in critically ill patients. Diagnosis is difficult with an inherent uncertainty and complicated by comorbidity, lack of routines for high-quality airway sampling and low sensitivity of routine microbiological tests. There is limited data on the aetiology and burden from HAP and VAP, and to the investigators knowledge, no previous prospective HAP and VAP studies has been performed in Norway. In the absence of rapid and accurate microbiological diagnosis, seriously ill HAP and VAP patients are often provided broad-spectrum antibiotics that have to be active on putative multi-drug resistant (MDR) bacteria, as failure to initiate prompt adequate therapy is associated with increased mortality. Overuse of broad-spectrum antibiotics promotes the selection and dissemination of MDR bacteria.

HVAPNOR brings together a multidisciplinary research team from Norwegian (Haukeland University Hospital (HUS), University of Bergen (UoB), Vestre Viken Hospital Trust (VVHF), and international institutions (Denmark, Netherlands and United Kingdom), with a strong record in respiratory disease research.

The overall aims of the HVAPNOR study are to improve diagnostic methods, antibiotic stewardship, treatment and management of HAP and VAP. The investigators will in a Norwegian context, map the incidence and the aetiology of HAP/VAP infections. During a two-year period, adult HAP and VAP patients admitted at HUS and VVHF, will be identified and voluntarily included in a prospective descriptive study. The project will strengthen the routines for adequate airway sampling and assess if provision of ultra-rapid, high-quality accurate molecular diagnostics will provide a more comprehensive microbiological etiological diagnose than routine analysis. A direct feedback to the clinician can facilitate pathogen-directed usage of antibiotics. We will evaluate the potential of molecular diagnostic platforms for the detection of pathogens and antimicrobial markers in HAP and VAP. Furthermore, the investigators will identify barriers that inhibit the acceptance of rapid molecular tests; and contribute to the optimisation of treatment protocols for HAP and VAP.

Finally, the study will also evaluate and identify new and clinically relevant diagnostic and prognostic biomarkers, including immune biomarkers and transcriptional profiling, in HAP and VAP.

The HVAPNOR study is in line with the objectives of the funding agencies, addresses clinical research activities to help to ensure that patients receive high-quality and reliable diagnostics and optimized treatment.

ELIGIBILITY:
A case definition of NV-HAP and VAP will be applied according to the 2005 American Thoracic Society and Infectious Disease Society of America´s clinical practice guidelines (unchanged in the 2016 revision).

Inclusion criteria:

* Age ≥18 years
* Meets case definition criteria (patient admitted to hospital or endotracheal intubation ≥ 48 hours, a new lung infiltrate + ≥2 of the following: temperature >38˚C, leukocytes <3.5 or >11.0, purulent secretions)
* Eligible for lower airways sampling
* Written informed consent

Exclusion criteria:

* Pulmonary embolism, segmental or larger
* Refractory septic shock (meeting the Sepsis-3 definition of septic shock, and requiring vasopressors ≥ 0.5 mcg/kg/min noradrenaline or equivalent dose of other vasopressor(s)
* Glasgow Coma Scale score 3
* Patients not eligible for lower airways sampling
* Palliative situation with life expectancy < 1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients developing pneumonia during hospital stay for other cause.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to microbiological diagnose | September 2020-August 2022
  Hours
Microbiological diagnose | September 2020-August 2022
  Microbes
Prevalence of resistance mutations | September 2020-August 2022
  Types and numbers
Change from empirical to targeted antimicrobial treatment | September 2020-August 2022
  Percentage based upon optimized microbiological diagnostics
Time to targeted antimicrobial treatment | September 2020-August 2022
  Hours

CONTACTS AND LOCATIONS:
Overall Officials: Lars Heggelund, MD, PhD, Principal Investigator — Vestre Viken Hospital Trust; Harleen Grewal, MD, PhD, Study Director — University of Bergen; Elling Ulvestad, MD, PhD, Study Director — University of Bergen
Locations (1):
- Vestre Viken Health Trust, Drammen, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, SAP and ICF will be made avialbe after the study has been initiated. CSR will be made avialbel after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: September 2020-December 2024.
Access Criteria: PI must be contacted